CLINICAL TRIAL: NCT00380419
Title: Infant Outcomes and Depression Treatment in Pregnancy
Brief Title: Effects of Interpersonal Psychotherapy on Depression During and After Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sheila M Marcus, Section Director Child & Adolescent Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00007344; R21MH072673 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Depression; Anxiety Disorders
Keywords: Pregnancy; Postpartum Depression
MeSH Terms: conditions — Depression; Anxiety Disorders; Depression, Postpartum | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive 16 sessions of interpersonal psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy (IPT)

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy (IPT) — IPT sessions will address adjustment to pregnancy, concerns about interpersonal relationships, and parenting concerns. Sessions will be weekly, but may be determined by clinical desires of patient and therapist.

SUMMARY:
This study will evaluate the impact of interpersonal psychotherapy on the course of depression during and after pregnancy, as well as its effect on infant birth outcomes.

DETAILED DESCRIPTION:
Depression is a serious illness that affects a person's body, mood, and thoughts. Researchers believe that it is one of the most common complications during and after pregnancy. The following symptoms may be signs of depression during pregnancy: 2 or more weeks of depressed mood; decreased interest or pleasure in activities; change in appetite or sleep patterns; fatigue or decreased energy; difficulty concentrating; excessive feelings of guilt or worthlessness; thoughts of suicide; and extreme restlessness or irritability. Depression is difficult to diagnose during pregnancy because its symptoms are sometimes confused with those of pregnancy. If left untreated, depression during pregnancy may affect not only the mother, but also the baby. Specifically, the hormone changes brought on by depression may contribute to premature and low-birth-weight infants. Interpersonal psychotherapy (IPT) is a short-term talking therapy that has been proven to be effective in treating depression. This study will evaluate the impact of interpersonal psychotherapy on the course of depression during and after pregnancy, as well as its effect on infant birth outcomes.

This study is associated with a larger parent study. Participants in this open-label study may be recruited directly for this study or through the parent study. All participants will receive 16 sessions of IPT. Sessions will last approximately 50 minutes and will focus on achieving depression symptom remission by improving interpersonal functioning. The majority of IPT sessions will be held prior to delivery; up to four sessions may be held postpartum. No medication will be provided in this study, but women who are currently taking selective serotonin uptake inhibitors (SSRIs) at the time of study entry may continue taking their medication. Participants whose symptoms do not improve with IPT will be referred to their non-study physician for further evaluation, and may begin taking SSRI medication upon physician recommendation. The effects of both IPT and medication therapy will be considered when assessing outcomes. Study visits will occur at 28, 32, and 36 weeks gestation, as well as Weeks 1, 2, and 6, and Month 6 postpartum. Measurements will include cortisol levels, which will be obtained using a saliva sample, as well as depression symptom severity, which will be assessed at each IPT session. Blood samples will be taken as part of the parent study.

ELIGIBILITY:
Inclusion Criteria:

* No more than 28 weeks pregnant at the time of study entry
* History of depression or anxiety
* Current symptoms of distress
* Score of 9 or greater on the Edinburgh Postnatal Depression Scale (EPDS)
* English-speaking

Exclusion Criteria:

* Plans to move away from the area prior to giving birth
* Current use of steroids for medical conditions

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Mothers' depression symptom severity, as determined by the 17-item Hamilton Rating Scale for Depression (HAM-D 17) | Measured during pregnancy and the first 7 months after delivery
Infant birth outcomes | Measured during the first 7 months after delivery

SECONDARY OUTCOMES:
Biologic measures related to depression in both mothers and infants | Measured through 14 months fter delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Marcus, MD, Principal Investigator — Universitiy of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States